CLINICAL TRIAL: NCT06733480
Title: Innovating Physical Therapy: A Pilot Study on Band Connect's Impact on Compliance, Satisfaction, and Revenue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Band Connect (Unknown)
Responsible Party: Principal Investigator, Robert J. Gillespie, Vice Chair of Education, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20241277
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Tears; Anatomic Total Shoulder Arthroplasty; Reverse Total Shoulder Arthroplasty
Keywords: physical therapy compliance; home-based physical therapy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 Band Connect (Experimental): Patients in group 1 will be set up with the Band Connect platform and build their treatment plan at the first in-clinic visit.
  Interventions: Device: Band Connect
- Group 2 Standard Care (No Intervention): Group 2 will consist of retrospective chart review to as act a control group. Charts will be pulled from 1/1/2019-12/31/2023.

INTERVENTIONS:
Device: Band Connect — Band Connect provides a medical-grade and condition-specific platform that augments the clinician workflow by extending the in-clinic MSK rehabilitation experience into the patient's home - leading to higher quality personalized treatment and increased adherence with enhanced economics and reimbursement for the clinic.
  Arms: Group 1 Band Connect

SUMMARY:
Participants are being invited to take part in this research study because you will be undergoing total shoulder replacement or rotator cuff repair and will be participating in physical therapy rehabilitation following the procedure. The purpose of this research is to investigate the effectiveness of Band Connect, a connected health platform, in enhancing compliance with home exercise programs among patients undergoing physical therapy. This study aims to evaluate the implications of increased compliance on improving patient engagement and increasing satisfaction for both patients and clinicians. Additionally, the study will analyze the economic implications of implementing Band Connect's hybrid care model on driving increased revenue per patient.

ELIGIBILITY:
Inclusion Criteria:

* Age range: from 18 to 89 years old
* Surgery performed by Dr. Robert Gillespie and will be undergoing post-op physical therapy rehabilitation at University Hospitals
* Patients undergoing primary anatomic total shoulder shoulder arthroplasty (aTSA) or primary reverse total shoulder arthroplasty (rTSA)
* Patients undergoing primary rotator cuff repair
* Prescribed outpatient physical therapy for post-operative rehabilitation

Chart Review Inclusion Criteria:

* Age range: from 18 to 89 years old
* Surgery performed by Dr. Robert Gillespie who underwent post-op physical therapy rehabilitation at University Hospitals
* Patients who underwent primary anatomic total shoulder shoulder arthroplasty (aTSA) or primary reverse total shoulder arthroplasty (rTSA)
* Patients who underwent primary rotator cuff repair
* Prescribed outpatient physical therapy for post-operative rehabilitation

Exclusion Criteria:

* Patients undergoing hemiarthroplasty or revision TSA
* Patients undergoing revision rotator cuff repair
* TSA performed for proximal humerus fractures
* Length of stay in hospital following shoulder surgery greater than 3 days
* Shoulder injuries related to workers compensation or involved in any pending litigation
* Pregnant individuals

Chart Review Exclusion Criteria:

* Patients undergoing hemiarthroplasty or revision TSA
* Patients undergoing revision rotator cuff repair
* TSA performed for proximal humerus fractures
* Length of stay in hospital following shoulder surgery greater than 3 days
* Shoulder injuries related to workers compensation or involved in any pending litigation
* Pregnant individuals

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of physical therapy visits as measured by medical record review. | Up to 6 months
Number of home exercise programs completed as measured by medical record review. | Up to 6 months
Number of in clinic visits as measured by medical record review. | Up to 6 months
Number of patients who were able to return to work | Up to 6 months
  This will be asked as a Yes/No question
Time to return to work measured in weeks | Up to 6 months
Number of patients who returned to sports | Up to 6 months
  This will be asked as a Yes/No question
Change in pain as measured by the Visual Analog Scale | Baseline, 1 month, 3 months, 6 months
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Active range of motion measured in degrees | Up to 6 months
Passive range of motion measured in degrees | Up to 6 months
Strength will be measured on a scale of 0-5 | Up to 6 months
  Strength scale:
  * 0: no visible or palpable contraction
  * 1: visible or palpable contraction without motion
  * 2: full range of motion, gravity eliminated
  * 3: full range of motion against gravity
  * 4: full range of motion against gravity, moderate resistance
  * 5: full range of motion against gravity, maximal resistance
Patient satisfaction as measured by American Shoulder and Elbow Surgeons (ASES) Score | Up to 6 months
  Scored out of 100, with higher scores indicating greater satisfaction
Number of adverse events as measured by medical record review. | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gillespie, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No